CLINICAL TRIAL: NCT03051412
Title: Differences in Pain Sensitivity in Young Females With Longstanding Patellofemoral Pain, Recovered Females With a History of PFP, and Healthy Controls.
Brief Title: Pain Mechanisms in Young Adolescent Females With Longstanding Patellofemoral Pain
Status: Completed | Type: Observational
Sponsor: Aalborg University (Other)
Collaborators: Research Unit for General Practice in Aalborg (Other)
Responsible Party: Principal Investigator, Sinead Holden, Post- Doctoral Research Fellow, Aalborg University
Other Study IDs: N-20160058 (1)
Record Dates: First submitted 2017-02-09; First posted 2017-02-13 (Actual); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Patellofemoral Pain Syndrome; Pain
MeSH Terms: conditions — Patellofemoral Pain Syndrome; Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Current Patellofemoral Pain: This group has current patellofemoral pain
  Interventions: Other: No Intervention
- Recovered: This group has a previous history of patellofemoral pain, but currently self reports as recovered.
  Interventions: Other: No Intervention
- Control: This is a control group with no history of knee pain.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No intervention

SUMMARY:
Patellofemoral pain (PFP) is a highly prevalent musculoskeletal condition in adult females, which is associated with decreased quality of life and physical activity levels. PFP is highly persistent, with up to 50% of adolescents reporting persistent pain at both one and two year follow-ups. Previous research has demonstrated altered pain sensitivity in in older individuals with chronic pain, however, less is known about this in conditions such as PFP, which is common in younger populations. Additionally it is unknown if these characteristics return to similar values as healthy controls, when symptoms resolve.

The aim of this study will be to compare pain sensitivity in individuals with PFP, compared to those with a previous history of PFP who currently are pain-free, and a control group with no history of knee pain.

DETAILED DESCRIPTION:
Recently it has been demonstrated that females with longstanding PFP demonstrate increased pain sensitivity, or hyperalgesia in the peripheral nervous system and impaired conditioned pain modulation, which is representative of decreased descending control of pain in the central nervous system. This is commonly seen in older adults with chronic longstanding pain, such as knee OA.

Understanding the evolution of pain mechanisms during recovery may yield important insights into the highly recurrent nature of this condition. Self-reported recovery appears to be associated with increased pressure pain thresholds, in comparison to those with current PFP. However, it is unknown whether these characteristics, along with centrally mediated pain processing, ever return to 'normal', or to the same levels of those with no history of pain.

To examine this, the investigation will compare the three groups (PFP versus Recovered versus Control), on measures of pain sensitivity (as defined in the primary and secondary outcomes), to determine differences between groups.

Demographic data, regarding age, height and weight will be collected, as well as pain frequency (almost daily, several times per week, weekly, monthly, rarely, never), pain intensity (measured on numeric rating scale), Knee Injury and Osteoarthritis Outcome score, and spatial distribution of pain (using the Navigate pain application). The group that self report as recovered, will be asked to report when their symptoms resolved.

A subgroup analysis will be undertaken in the recovered group, to examine the relationship between the time since last knee pain was experienced, (duration they self- report being symptom-free), and pain sensitivity, as assessed by the primary and secondary outcome measures.

Participants will be recruited from the Adolescent Pain in Aalborg (APA2011) cohort. In 2011, a cohort of 2200 adolescents aged 15 to 19 years answered an online questionnaire on musculoskeletal pain. Of these, 504 reported knee pain, and 153 of these were clinically diagnosed with PFP. Five years later, the 504 adolescents, as well as 252 randomly selected adolescents who did not report knee pain in 2011, completed a follow-up questionnaire regarding current pain (clinical trials.gov identifier: NCT02873143). From this group, a sample of participants' who were diagnosed with PFP in 2011, and self report with current pain, or as 'recovered' will be randomly contacted for inclusion in the current investigation (PFP and recovered groups respectively). Additionally, of the control participants from the original APA2011 cohort, who reported no pain in 2011, and no pain in 2016, a random sample will be drawn and invited to participate as the control group.

If this cohort is insufficient to reach the required sample size (n = 36 in each group), participants will be recruited through other sources such as GP's, and social media.

Embedded within this cross-sectional study, is a randomized crossover trial (in the group with PFP) which has been approved by the local ethical committee under the same approval number (N-20160058). This can be accessed on clinicaltrials.gov under the title "The acute effects of hip and knee exercises on pain sensitivity in young adult females with long-standing patellofemoral pain - a randomized crossover study." with Dr. Michael Rathleff as the primary investigator.

ELIGIBILITY:
Patellofemoral Pain Group:

Inclusion:

* Female
* Age 18-30years
* Current longstanding patellofemoral pain

Exclusion Criteria:

* Patients who have sustained a traumatic injury to the hip, knee, ankle or the lumbar spine within the past 3 month will be excluded.
* Participants will be excluded if they have other diagnosable pathologies that can cause pain around the kneecap (patellatendinopathy, Osgood-Shlatter, iliotibial band syndrome, Sinding-Larsen-Johansson syndrome, reverse jumper) if they occur in isolation (without patellofemoral pain).

Recovered Group:

Inclusion:

* Previous history of patellofemoral pain, reporting no current knee pain
* Female
* Aged 18-30 years

Exclusion:

* Participants will be excluded if they have other diagnosable pathologies that can cause pain around the kneecap (patellatendinopathi, Osgood-Shlatter, iliotibial band syndrome, Sinding-Larsen-Johansson syndrome, reverse jumper)
* Other pain conditions

Control:

Inclusion:

* Female
* Aged 18-30

Exclusion:

* Current knee or other other musculoskeletal pain
* Previous history of knee or musculoskeletal pain

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population will consist of young females. One group will include participants with current longstanding patellofemoral pain, while a second group will include those with a history of pain, who self report as recovered, and a control group, who has no previous history of knee pain.
Sampling Method: Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2017-02-22 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Conditioned pain modulation | Baseline
  Conditioned pain modulation (CPM) will be assessed using cuff algometry

SECONDARY OUTCOMES:
Pressure pain thresholds will be measured around the lower leg and forearm | baseline
  Mechanical pressure pain thresholds will be assessed using a handheld algometer to assess distal and remote hyperalgesia.
Pressure Pain thresholds at the knee | baseline
  Mechanical pressure pain thresholds will be assessed using a handheld algometer to assess local hyperalgesia.
Temporal summation of pain | baseline
  Temporal summation is be induced by 10 short-lasting stimuli (1 sec each) at the level of PTT given with a 1 sec break in between stimuli using the cuff algometry. Subject will be instructed to rate the pain intensity after each stimulus using an electronic VAS scale.
Pressure detection & pressure tolerance threshold assessed by cuff algometry | baseline
  Pressure detection & tolerance thresholds will be assessed bilaterally on the lower extremity using cuff algometer.

CONTACTS AND LOCATIONS:
Overall Officials: Sinead Holden, PhD, Principal Investigator — Research Unit for General Practice, Department of Clinical Medicine, Aalborg University
Locations (1):
- Research Unit for General Practice in Aalborg, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: Undecided